CLINICAL TRIAL: NCT06066463
Title: My Skin & Hair Journey_virtual Registry
Status: Suspended | Type: Observational
Why Stopped: recruitment issue
Sponsor: L'Oreal (Industry)
Collaborators: Verily Life Sciences (Unknown)
Responsible Party: Sponsor
Other Study IDs: ACR/MYSH/23-05335
Record Dates: First submitted 2023-09-27; First posted 2023-10-04 (Actual); Last update posted 2025-11-03 (Actual); Status verified 2025-10

CONDITIONS: Skin; Hair
MeSH Terms: interventions — Surveys and Questionnaires

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Patient Registry: Yes
Target Follow-Up Duration: 18 Months
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

INTERVENTIONS:
Behavioral: questionnaires — Self reported female gender

SUMMARY:
This is a longitudinal, observational, direct to participant registry to better understand biological, clinical, and environmental aspects of skin/hair health and beauty.

DETAILED DESCRIPTION:
This is a longitudinal, observational, direct to participant registry to better understand biological, clinical, and environmental aspects of skin/hair health and beauty. By collecting, organizing, and analyzing data for a group of participants over time, researchers will use information to learn more about these topics. This study will collect long-term information about study participants, developing a lean, participant-centric approach to curating meaningful longitudinal data that incorporate participant perspectives including quality of life and personal beauty health preferences. This should allow researchers to understand how participant skin health changes over time and what factors can inﬂuence those changes with a speciﬁc focus on participant-centric learning.

Additionally, this study will look for ways to develop and/or improve data handling approaches to increase the depth, generalizability, and/or longitudinality of skin health and beauty data based on approaches that decrease burden, as appropriate, over time (eg, for study participants, investigators, clinical research stakeholders)

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to provide informed consent
* Willing and able to provide applicable privacy authorization(s)
* Current resident of the United States
* 18 to 70 years of age at the time of informed consent Self identiﬁed female gender
* Able to read and understand English and/or Spanish
* Ability to access internet based study-related tools (eg, applications, software, email notiﬁcations)
* Willingness to use study web/mobile applications (eg, selﬁe assistant, air quality and weather monitoring)

Exclusion Criteria:

- Employee of the Sponsor(s), contracted research organizations, or virtual research sites

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Gender Based: Yes — self declare women
Study Population: healthy Female self declared
Sampling Method: Non-Probability Sample
Enrollment: 10000 (Estimated)
Dates: Start 2023-06-30 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2025-11-30 (Estimated)

PRIMARY OUTCOMES:
Collect and organize a longitudinal skin & hair beauty registry | 18 months
  Collect and organize a longitudinal skin & hair beauty registry that links skin & hair individual outcomes to lifestyle, environment, age and beauty perception on all skin diversity, and to make that information accessible and actionable for researchers and consumers.

SECONDARY OUTCOMES:
Build and improve generalizable beauty knowledge | 18 months
  Build and improve the broader longitudinal registry from various data sources inclusive of intentionally collected data and other supporting data to inform generalizable beauty knowledge
improve insights from longitudinal data | 18 months
  Support the development and/or optimization of people, process, and technical approaches to improve insights from longitudinal data (eg, to improve research approaches, guide advances in precision beauty)

CONTACTS AND LOCATIONS:
Overall Officials: KRISDA CHAIYACHATI, MD MPH FACP, Principal Investigator — Verily Life Sciences
Locations (1):
- Verily Life Sciences, South San Francisco, California, United States

IPD SHARING:
Plan to Share IPD: No